CLINICAL TRIAL: NCT06104085
Title: 99mTc-MY6349 SPECT/CT Imaging in Trop2-positive Triple-negative Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K4429
Record Dates: First submitted 2023-09-03; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-MY6349 SPECT/CT (Experimental): Inject 99mTc-MY6349 and then perform SPECT/CT scan.
  Interventions: Diagnostic Test: 99mTc-MY6349 SPECT/CT scan

INTERVENTIONS:
Diagnostic Test: 99mTc-MY6349 SPECT/CT scan — Triple-negative breast cancer patients underwent 99mTc-MY6349 SPECT/CT imaging to observe the binding ability of this tracer to Trop2 in the tumor and the uptake of the drug by the tumor, combined with the pathological expression level of Trop2 in the patient's lesions and 18F-FDG PET/CT imaging uptake to evaluate the efficacy of 99mTc-MY6349 in the diagnosis of triple-negative breast cancer; at the same time, combined with the treatment effect of patients using the anti-Trop2 targeted antibody gosatuzumab, the analysis of 99mTc-MY6349 SPECT/CT imaging prediction of prognosis in patients with triple-negative breast cancer treated with gosatuzumab.

SUMMARY:
Human trophoblast cell-surface glycoprotein antigen 2 (Trop2) is a membrane surface receptor that plays an important role in the occurrence and development of tumors. Studies have shown that Trop2 is highly expressed in a variety of cancers (such as breast cancer, lung cancer, gastric cancer, colorectal cancer, pancreatic cancer, prostate cancer, cervical cancer, head and neck cancer, and ovarian cancer, etc.) and is related to the proliferation, invasion, and metastasis of tumor cells. and other processes related. According to statistics, more than 80% of breast cancer patients highly express Trop2, and high expression of Trop2 is positively correlated with shortened survival and poor prognosis of cancer patients. In this study, a single-domain antibody targeting Trop2 was selected to prepare a new nuclear medicine molecular probe 99mTc-MY6349, so as to monitor the expression level of Trop2 in patients' systemic tumors through SPECT/CT imaging. Breast cancer patients who intend to use gosatuzumab for subsequent treatment can first undergo 99mTc-MY6349 SPECT/CT imaging to detect Trop2 expression levels in systemic tumors. Subsequently, 18F-FDG PET/CT imaging was performed to compare and detect the distribution of primary tumors and systemic metastases in patients with breast cancer. This study analyzes the heterogeneity of Trop2 expression levels within the primary tumor and the heterogeneity of expression levels in systemic metastases, thereby providing a basis for testing whether the patient is suitable for subsequent treatment and conducive to the formulation of subsequent treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged between 18 and 80 years old.
* Patients with suspected or definite diagnosis of triple-negative breast cancer.
* Patients with suspected or confirmed triple-negative recurrent or metastatic breast cancer.
* Female subjects must have medical records to prove that they have undergone surgical sterilization (such as hysterectomy, bilateral oophorectomy, or tubal ligation) or have been menopausal for more than one year; if they still have the ability to conceive, isolation contraceptive measures must be taken during this study period.

Exclusion Criteria:

* Suffering from severe gastrointestinal, cardiovascular, liver, kidney, blood system, endocrine, respiratory system, immune deficiency and other serious diseases.
* Claustrophobia.
* In the past year, due to other clinical medical treatment or scientific research needs, received ionizing radiation outside the scope of this experiment, so that the annual radiation exposure dose exceeded 50mSv.
* Pregnant or lactating women.
* Received experimental drug or device treatment (with unclear efficacy or safety) within 1 month.
* There is any situation in which the conductor of this study believes that any aspect related to this experiment may cause harm or be potentially harmful.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
semi-quantitative analysis | through study completion, an average of 1 year
  use the region of interest (ROI) method to measure the ratio of uptake at the lesion site to liver uptake

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China